CLINICAL TRIAL: NCT06361043
Title: Conebeam CT-based Online Adaptive Radio-Therapy for Esophageal Cancer (ARTEC)
Acronym: ARTEC
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01833
Record Dates: First submitted 2024-03-25; First posted 2024-04-11 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite multimodal therapy, patients with esophageal cancer have poor prognosis with 5-year overall survival around 25%. Considering tumor-related death as main reason for high mortality rate in those patients, treatment-related cardio-pulmonary toxicities could also play a role in this regard. Online adaptive radiotherapy offers the possibility for daily re-planning and therefore helps radiation oncologists to better spare the organs at risk and reduce radiation-induced toxicity. Tha aim of ARTEC is to assess the pulmonary toxicity in patients with esophageal cancer treated with online adaptive radiotherapy.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is currently the tenth most common cancer and sixth leading cause of cancer-related mortality worldwide. Multimodal treatment strategy consisting of surgery with pre-/perioperative Radio-/chemotherapy (RCHT) regimens the standard of care for non-metastatic locally advanced EC. However, the treatment of EC is challenging and the risk of tumor recurrence remains high. Furthermore, toxicities of such combined treatments can be substantial and there is room for optimization of RT to reduce the radiation dose to heart and lungs. While 3D-conformal radiotherapy is traditionally used for treatment of EC, modern irradiation techniques, such as intensity-modulated radiotherapy (IMRT) or volumetric intensity modulated arc therapy (VMAT), are increasingly implemented in the management of EC. The investigators know from literature that esophageal motion could be a challenge and therefore bigger margins are needed to achieve an acceptable tumor coverage. In addition to positioning and motion uncertainties, there could be a substantial inter-fractional tumor size reduction during RCHT. Tumor shrinkage can consequently lead to OARs shifting into the target volumes, which results in excess radiation dose to OARs with increased toxicity. Adaptive radiotherapy (ART) is a treatment technique to do a re-planning during the course of treatment to adjust the delivery of radiation dose based on geometrical changes of tumor and OARs. Considering the uncertainties in OAR and tumor displacement positioning, as well as tumor size reduction during RCHT, makes EC a perfect candidate for ART. This single-arm prospective study aims to assess pulmonary toxicity and dosimetrical analysis of ART for EC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed diagnosis of AC (Adenocarcinoma) or SCC (squamos cell carcinoma) of the thoracic esophagus or gastroesophageal junction (Siewert I-II)
* Patients with cT2-4b cN0 cM0 or cTany cN+ cM0 or any patient with early stage EC ineligible for upfront surgery
* Age >= 18 years old
* Karnofsky Performance Status (KPS) >= 70 or ECOG (Eastern Cooperative Oncology Group) 0 - 1
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with patients before registration in the trial

Exclusion Criteria:

* Cervical esophageal cancers (15-18 cm from the incisors)
* Definitive clinical or radiologic evidence of metastatic disease
* Any active malignancy within 2 years of study registration that may alter the course of esophageal cancer treatment
* Prior thoracic radiotherapy that would result in overlap of radiation therapy fields
* Induction chemotherapy for the current malignancy prior to RCHT is allowed if last dose is no more than 90 days and no less than 10 days prior to registration
* Pregnant and/or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal cancer (EC) is currently the tenth most common cancer and sixth leading cause of cancer-related mortality worldwide. Multimodal treatment strategy consisting of surgery with perioperative chemotherapy or preoperative radio-chemotherapy (RCHT) regimens the standard of care for locally advanced and potentially curable EC. For patients who decline surgery or patients in poor general condition and unfit for tumor resection, definitive RCHT alone could be considered as a reasonable treatment option.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pulmonary toxicity | Up to 12 months after RCT
  The primary endpoint of this prospective study is pulmonary toxicity after concurrent radio-chemotherapy for patients with esophageal cancer treated with ART. According to literature, around 10 - 25%- of EC patients experience radiation induced pulmonary complications (RIPC) after combined radio-chemotherapy. However, the high rates of toxicity (up to 25%) were seen in patients irradiated with old RT techniques, such as 3D-CRT (Conformal Radiotherapy). New data, using modern RT, show much less pulmonary toxicity (10%). RIPC includes mostly radiation pneumonitis, radiation pulmonary fibrosis and pleural effusion .

SECONDARY OUTCOMES:
Number of patients with pathological complete response | Directly after surgery up to two weeks
  A pathological complete response (pCR) is defined as the lack of all signs of cancer in tissue samples removed during surgery or biopsy after treatment with RCHT. To find out if there is a pCR, a pathologist checks the tissue samples to see if there are still cancer cells left after the anticancer treatment.
Dosimetrical analysis between scheduled and adaptive plans | Directly after radiotherapy up to two weeks
  Dosimetrical analysis between scheduled and adaptive plans.
  We set the dosimetric goals for target volumes and OARs as follows:
  * CTV coverage: D95% >= 100.0%*
  * PTV coverage: D95% >= 100.0%
  * PTV Dminimum: D99% >= 99.0%
  * PTV Dmaximum: D1.0% <= 101.0%
  * Heart: Dmean < 18Gy°
  * Lung: V20Gy < 20% and mean lung dose (MLD) < 12Gy - Liver: Dmean < 18Gy"
    * Dose that covers 95% of target volume is equal or more than 100% of prescribed dose.
  "Mean Dose to the heart should be less than 18Gy "Mean dose to the liver should be less than 18Gy
  All these values will be extracted from treatment planning system (TPS) for both adaptive and scheduled plans. Comparing these two data sets, we will demonstrate if patients profited from OART from dosimetrical point of view

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Hemmatazad, MD, Study Chair — Inselspital Bern, Department of Radio-Oncology
Locations (1):
- Inselspital, University of Berne, Deparftment of Radio-Oncology, Bern, Switzerland